CLINICAL TRIAL: NCT05549830
Title: The Effect of Different Positioning Before, During and After Surgery on Pressure Injury: a Randomized Controlled Study Protocol
Brief Title: Effect of Different Positioning Before, During and After Surgery on Pressure Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MarmaraU_bedia_guler
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Pressure Injury; Injuries
Keywords: Surgical pressure injury; Prevention; Patient positioning
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries | interventions — Patient Positioning; Postoperative Period

STUDY DESIGN:
Intervention Model Description: In this trial, a two-group design will be used, with an equal number of random participants assigned to each group
Masking Description: Masking will not be used. Participants meeting the inclusion criteria will be assigned to one of the two groups by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): During the night before surgery and for the first 36 hours after surgery, the participants assigned to the intervention group will be placed in positions different from surgical positions.
  After surgery the patient will be placed in a different position compared to during surgery, with repositioning being undertaken every two hours until the first 36th postoperative hour, and the development of pressure injuries will be evaluated at the 36th hour. If no pressure injury has developed in this period, the patient will be placed in the surgical position for a duration that will not exceed 30 minutes, and then repositioning will be applied at two-hour intervals. If pressure injuries have developed, different repositioning techniques will continue to be applied at two-hour intervals.
  Interventions: Other: Patient Positioning
- Control Group (No Intervention): The control group will only receive routine care. The positions of the patients in this group will be monitored and recorded at two-hour intervals.

INTERVENTIONS:
Other: Patient Positioning — In the preoperative period, the patient/patient relative will be informed about the possible surgical position and the importance of placing the patient in a different position before and after surgery.
  İn the postoperative period, the patient will be placed in a different position compared to during surgery, with repositioning being undertaken every two hours until the first 36th postoperative hour, and the development of pressure injuries will be evaluated at the 36th hour. If no pressure injury has developed in this period, the patient will be placed in the surgical position for a duration that will not exceed 30 minutes, and then repositioning will be applied at two-hour intervals. If pressure injuries have developed, different repositioning techniques will continue to be applied at two-hour intervals.
  Other Names: Place the patient in a different position compared to during surgery, In the preoperative and postoperative periods.
  Arms: Intervention Group

SUMMARY:
Background: Patients undergoing surgery are at risk of developing pressure injuries since they remain in a fixed position on the operating table under anesthesia for a long time. In the management of surgical patients, the prevention of surgical pressure injuries is the best strategy, requiring effective risk assessment and timely implementation of preventive interventions.

Aim: To evaluate the effect of preoperative and postoperative patient repositioning other than intraoperative positions on the development of pressure injuries.

H1 Hypothesis: In the preoperative and postoperative periods, there is a significant difference in the development of pressure injuries between patients who have been repositioned using non-surgical positions compared to those that did not undergo this intervention.

Methods: This study has been designed as a prospective randomized controlled trial. Patients meeting the inclusion criteria of the trial will be allocated to the intervention and control groups using a random number generator. The participants to be assigned to the intervention group will be placed in different positions other than their surgical positions on the night before surgery and until the first 36 hours after the operation, while the control group will only receive routine care. The groups will be evaluated in terms of pressure injury development for at least 72 hours until the end of the postoperative sixth day or discharge from the hospital.

DETAILED DESCRIPTION:
INTRODUCTION

Surgical interventions constitute one of the many risk factors that cause the development of pressure injuries. Since patients are in an immobile and fixed position during surgery and under the effect of anesthetic agents, they cannot feel the pain caused by pressure and shear forces or change their positions.Therefore, all patients undergoing surgical interventions are at risk of developing pressure injuries.

Surgical pressure injuries are those that occur during surgery or within the first 72 hours or first six days after surgery, and they are considered to be important complications that can have undesirable consequences. The development of surgical pressure injuries not only increases postoperative recovery time and length of hospital stay but also results in additional treatment requirement and pain experience for the patient, have adverse physical, mental, and financial effects, poses a risk of infection, and leads to reduced quality of life and deformities. In addition, the perioperative development of these injuries is an important indicator of the quality of care in terms of both the patient and the healthcare center and a serious safety issue for the former.

Despite technological advances, surgical pressure injuries remain a clinical problem for patients undergoing surgery. According to national and international studies, the prevalence of these injuries ranges from 0.3% to 66%, accounting for 4% to 45% of all hospital-acquired pressure injuries and shows an increasing trend in recent years. Among the risky surgical interventions listed in the literature are cardiac, general (abdominal and hepatobiliary), orthopedic, neurosurgical, vascular, urological, and thoracic operations.

The best strategy to manage pressure injuries is prevention rather than treatment. In this regard, it is recommended to perform an effective risk assessment and implement timely preventive interventions. The primary step is risk assessment, including the evaluation of associated risk factors and a comprehensive examination of skin condition, which helps identify high-risk cases in which to implement preventive interventions. Although many risk factors have been reported to contribute to the development of pressure injuries in patients undergoing surgery, the most important evidence-based risk factors have been shown to be preoperative immobility time, operation time, intraoperative hypothermia and hypotension, and immobility on the first postoperative day (level of evidence: weak; strength of recommendation: strong). Recommendations for prevention include patient positioning in a way to reduce the risk of pressure injury development during surgery (level of evidence: weak; strength of recommendation: strong), use of pressure support surfaces on the operating table (level of evidence: strong; strength of recommendation: weak), and redistribution of pressure before and after surgery (level of evidence: weak; strength of recommendation: strong). It is recommended that patients should be placed in different positions before and after surgery to redistribute pressure. However, there are a limited number of studies in the literature investigating the effectiveness of this application, which is based on a weak level of evidence but a strong recommendation, and it is emphasized that there is a need for further studies focusing on post-anesthesia nursing care and standards in practice.

Patient positioning plays a key role in the prevention of pressure injuries, and repositioning is recommended in all patients at risk of developing these injuries unless contraindicated (level of evidence: strong; strength of recommendation: strong). Patient repositioning aims to reduce the duration and size of pressure over bony prominences and increase the duration of the resistance of tissues. This is a cost-free, non-invasive, and effective method of redistributing pressure. In a study investigating the effect of a postoperative care bundle that included placing the patient in different positions other than those used during surgery, prophylactic dressing applied at pressure points, and use of an intraoperative pressure support surface, it was reported that the incidence of pressure injuries in the patients was completely eliminated at the end of the second year.

Considering the suggestion that placing the patient in a position different from surgical positions as long as possible will help distribute the pressure to other pressure points, thus shortening the length of time during which the tissue is at risk and reducing the risk of developing pressure injuries, we have designed the current study to investigate the effects of preoperatively and postoperatively repositioning patients on the development of pressure injuries.

METHODS

Trial design:

In this trial, a two-group design will be used, with an equal number of random participants assigned to each group.

Setting:

The trial will be carried out at the general surgery clinic and intensive care unit (ICU) of a training and research hospital in Bursa, Turkey.

Participants and sampling:

The sample of the study was determined with the power analysis using G*Power 3 (2007) software. Based on the pressure injury rates reported on the first postoperative day for the patient groups included in the study of Guo et al. (17.65% in the control group, 0% in the intervention group), the effect size (d) was calculated as 0.31 to achieve a statistical test power (1-β) of 80% at a type I error (α) of 0.05, and taking into account the standard deviation value, the minimum number of participants to be included in the sample was determined as 88 (44 for each group). However, we decided to include a total of 100 patients (50 in the intervention group and 50 in the control group) in order to prevent a decrease in test power due to the possibility of data loss during data collection.

Randomization:

The participants will be determined from the surgery list, and those meeting the inclusion criteria will be randomly assigned to either group using a random number generator (https://www.randomizer.org).

Instruments:

Study data will be collected using an individual and clinical characteristics form, the Munro Pressure Ulcer Risk Assessment Scale (Munro scale), the Patient Mobility and Observer Mobility Scale, a pressure injury diagnosis and staging form, and a patient follow-up form.

Ethical considerations:

For the collection of study data, ethical approval was obtained from the Clinical Research Ethics Committee of Uludag University Faculty of Medicine (decision number: 2022-4/36, date: 23.02.2022) and written permission from the institution where the study will be conducted. In addition, for the scales to be used in the study, written permission was received from the authors who performed their validity and reliability analyses in Turkey. During the data collection process, informed voluntary verbal and written consent will be obtained from all the participants after explaining the purpose of the research, study procedure, and their rights in this process. Throughout the study, we will follow the principles of the Declaration of Helsinki 2008 and Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Being scheduled to undergo elective major abdominal surgery that is expected to take three or more hours,
* Being aged 18 years or older,
* Having no communication problems,
* Being able to communicate in Turkish,
* Being conscious and having intact orientation function, i.e., awareness of place, person, and time,
* Providing written informed consent to participate in the study.

Exclusion Criteria:

* Being planned to undergo emergency major abdominal surgery,
* Having preoperative pressure injuries.

Exclusion Criteria to be Applied After the İnitiation of the Study:

* Defined as developing a contraindicated condition during postoperative positioning,
* Being discharged within the first 72 hours postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Surgical pressure injury development | From at least 72 hours after surgery until the sixth postoperative day or discharge from the hospital if earlier.
  Surgical pressure injuries will be assessed in six categories: stage I, non-blanchable erythema; stage II, partial-thickness skin loss; stage III, full-thickness skin loss; stage IV, full-thickness tissue loss; unstageable, depth unknown; and suspected deep tissue injury, depth unknown, according to the international classification system included in the "Prevention and Treatment of Pressure Ulcers: Quick reference Guide, 2014" published by the National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel, and Pan Pacific Pressure Injury Alliance (NPUAP/EPUAP/PPPIA).

CONTACTS AND LOCATIONS:
Overall Officials: Bedia Güler, Nurse, Principal Investigator — Marmara University, Institute of Health Sciences
Locations (1):
- Marmara University, Institute of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walton-Geer PS. Prevention of pressure ulcers in the surgical patient. AORN J. 2009 Mar;89(3):538-48; quiz 549-51. doi: 10.1016/j.aorn.2008.12.022. PMID 19269379
- [Background] National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel and Pan Pacific Pressure Injury Alliance (NPUAP/EPUAP/PPPIA). Prevention and Treatment of Pressure Ulcers: Quick Reference Guide. Emily Haesler (Ed.). Cambridge Media: Perth, Australia; 2014.
- [Background] Shafipour V, Ramezanpour E, Gorji MA, Moosazadeh M. Prevalence of postoperative pressure ulcer: A systematic review and meta-analysis. Electron Physician. 2016 Nov 25;8(11):3170-3176. doi: 10.19082/3170. eCollection 2016 Nov. PMID 28070249
- [Background] Peixoto CA, Ferreira MBG, Felix MMDS, Pires PDS, Barichello E, Barbosa MH. Risk assessment for perioperative pressure injuries. Rev Lat Am Enfermagem. 2019 Jan 17;27:e3117. doi: 10.1590/1518-8345.2677-3117. PMID 30698218
- [Background] Spruce L. Back to Basics: Preventing Perioperative Pressure Injuries. AORN J. 2017 Jan;105(1):92-99. doi: 10.1016/j.aorn.2016.10.018. PMID 28034406
- [Background] Primiano M, Friend M, McClure C, Nardi S, Fix L, Schafer M, Savochka K, McNett M. Pressure ulcer prevalence and risk factors during prolonged surgical procedures. AORN J. 2011 Dec;94(6):555-66. doi: 10.1016/j.aorn.2011.03.014. PMID 22118201
- [Background] Munro CA. The development of a pressure ulcer risk-assessment scale for perioperative patients. AORN J. 2010 Sep;92(3):272-87. doi: 10.1016/j.aorn.2009.09.035. PMID 20816101
- [Background] Kandemir D, Yüksel S. Effective evidence-based interventions in preventing surgical pressure injuries. Journal of Hacettepe University Faculty of Nursing. 2021;8(1):85-92.
- [Background] Buso FD, Ferreira MB, Felix MM, Galvão CM, Barichello E, Barbosa MH. Pressure injury related to surgical positioning and associated factors. Acta Paul Enferm. 2021;34:eAPE00642.
- [Background] Ramezanpour E, Emami ZA, Heidari MA, Yazdani CJ, Moosazadeh M, Shafipour V. Incidence and risk factors of pressure ulcers among general surgery patients. Journal of Nursing and Midwifery Sciences. 2018;5(4 ).
- [Background] Kim JM, Lee H, Ha T, Na S. Perioperative factors associated with pressure ulcer development after major surgery. Korean J Anesthesiol. 2018 Feb;71(1):48-56. doi: 10.4097/kjae.2018.71.1.48. Epub 2017 Jul 4. PMID 29441175
- [Background] Chen Y, He L, Qu W, Zhang C. Predictors of Intraoperative Pressure Injury in Patients Undergoing Major Hepatobiliary Surgery. J Wound Ostomy Continence Nurs. 2017 Sep/Oct;44(5):445-449. doi: 10.1097/WON.0000000000000356. PMID 28877110
- [Background] Shaw LF, Chang PC, Lee JF, Kung HY, Tung TH. Incidence and predicted risk factors of pressure ulcers in surgical patients: experience at a medical center in Taipei, Taiwan. Biomed Res Int. 2014;2014:416896. doi: 10.1155/2014/416896. Epub 2014 Jun 26. PMID 25057484
- [Background] Guo Y, Zhao K, Zhao T, Li Y, Yu Y, Kuang W. The effectiveness of curvilinear supine position on the incidence of pressure injuries and interface pressure among surgical patients. J Tissue Viability. 2019 May;28(2):81-86. doi: 10.1016/j.jtv.2019.02.005. Epub 2019 Feb 25. PMID 30878174
- [Background] Akan C, Sayın YY. Prevalence of pressure injuries and risk factors in long-term surgical procedures. Bezmialem Science. 2021;9(1):75-83
- [Background] Karadag M, Gumuskaya N. The incidence of pressure ulcers in surgical patients: a sample hospital in Turkey. J Clin Nurs. 2006 Apr;15(4):413-21. doi: 10.1111/j.1365-2702.2006.01369.x. PMID 16553754
- [Background] Gurkan A, Kirtil I, Aydin YD, Kutuk G. Pressure injuries in surgical patients: a comparison of Norton, Braden and Waterlow risk assessment scales. J Wound Care. 2022 Feb 2;31(2):170-177. doi: 10.12968/jowc.2022.31.2.170. PMID 35148625
- [Background] Black J, Fawcett D, Scott S. Ten top tips: preventing pressure ulcers in the surgical patient. Wounds International. 2014;5(4).
- [Background] Chen HL, Chen XY, Wu J. The incidence of pressure ulcers in surgical patients of the last 5 years: a systematic review. Wounds. 2012 Sep;24(9):234-41. PMID 25874704
- [Background] Scott SM. Progress and Challenges in Perioperative Pressure Ulcer Prevention. J Wound Ostomy Continence Nurs. 2015 Sep-Oct;42(5):480-5. doi: 10.1097/WON.0000000000000161. No abstract available. PMID 26336045
- [Background] Lumbley JL, Ali SA, Tchokouani LS. Retrospective review of predisposing factors for intraoperative pressure ulcer development. J Clin Anesth. 2014 Aug;26(5):368-74. doi: 10.1016/j.jclinane.2014.01.012. Epub 2014 Aug 10. PMID 25113424
- [Background] Haisley M, Sorensen JA, Sollie M. Postoperative pressure injuries in adults having surgery under general anaesthesia: systematic review of perioperative risk factors. Br J Surg. 2020 Mar;107(4):338-347. doi: 10.1002/bjs.11448. Epub 2020 Jan 21. PMID 31960958
- [Background] Walsh M. Pressure ulcer prevention. AORN J. 2011 Feb;93(2):197-8. doi: 10.1016/j.aorn.2010.12.012. No abstract available. PMID 21281759
- [Background] Kimsey DB. A Change in Focus: Shifting From Treatment to Prevention of Perioperative Pressure Injuries. AORN J. 2019 Oct;110(4):379-393. doi: 10.1002/aorn.12806. PMID 31560439
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343